CLINICAL TRIAL: NCT00126815
Title: Mathematical Modeling Analysis of Serum Prostate Specific Antigen After Radiotherapy
Status: Completed | Type: Observational
Sponsor: AHS Cancer Control Alberta (Other)
Collaborators: Cross Cancer Institute (Other)
Responsible Party: Sponsor
Other Study IDs: NA-15-0002
Record Dates: First submitted 2005-08-03; First posted 2005-08-05 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2011-12

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; prostate specific antigen; radiotherapy; mathematical modeling
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Clinical data are being used to build a mathematical model to describe the clinical results of radiotherapy for prostate cancer.

DETAILED DESCRIPTION:
Clinical data (prostate-specific antigen [PSA] response after radiotherapy) are being used to build a mathematical model to describe the clinical results of radiotherapy for prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Prostate cancer treated with radiotherapy +/- hormones

Exclusion Criteria:

* Prostatectomy

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2004-02; Primary Completion 2008-03 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Parliament, MD, Principal Investigator — AHS Cancer Control Alberta
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada